CLINICAL TRIAL: NCT01042223
Title: Laryngomalacia Exposed
Status: Completed | Type: Observational
Sponsor: Boushahri Clinic Medical Center (Other)
Responsible Party: Principal Investigator, Mohamed Said El-Sayed, Professor, Boushahri Clinic Medical Center
Other Study IDs: Boushahri Clinic
Record Dates: First submitted 2008-12-01; First posted 2010-01-05 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Complications
Keywords: Factors Predisposing or Causing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Laryngomalacia is the most common congenital laryngeal anomaly and the most frequent cause of stridor in infants and children. Symptoms usually appear within the first 2 weeks of life. Its severity increases up to 6 months. 15-60% of infants with laryngomalacia have synchronous airway anomalies.

DETAILED DESCRIPTION:
The most common health complications associated with laryngomalacia were: 1. Gastroesophageal reflux which was presented by arching, choking, gagging, feeding aversion and continuous crying 2. Frequent unilateral eye infections 3. Repeated choking, frequent vomiting and poor weight gain 4. Repeated upper respiratory tract infections (viral and bacterial), coughing and cyanosis 5. Repeated secretory otitis media 6. Aspiration pneumonia

ELIGIBILITY:
Inclusion Criteria:

* 500 full term babies ≥ 37 weeks of both sexes were delivered by different modes of delivery, with birth weights of ≥ 2.5 kg, with no history of natal complications and from the same community.
* Mothers of these babies are from different socioeconomic standards with different educational levels.

Ages: 14 Days to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinics
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S EL-Sayed, MBBCh, MSc, MD, Principal Investigator — New Children's Hospital, Cairo University
Locations (1):
- Boushahri Clinic Medical Center, Kuwait City, P.O.Box :698 Salmiya, Kuwait